CLINICAL TRIAL: NCT03760965
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin as Monotherapy in Chinese Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Diet and Exercise
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo in Chinese Patients With Type 2 Diabetes Mellitus Not Adequately Controlled by Diet and Exercise
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sanofi ended collaboration with Lexicon for Sotagliflozin. In China no regulatory pathway to transfer sponsorship during the conduct of ongoing studies.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC15194; U1111-1195-6181 (Other: UTN)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sotagliflozin dose 1 (Experimental): Sotagliflozin dose 1, given as two (2) dose 2 tablets, once daily, before the first meal of the day
  Interventions: Drug: sotagliflozin (SAR439954)
- Sotagliflozin dose 2 (Experimental): Sotagliflozin dose 2, given as 1 sotagliflozin dose 2 tablet and 1 sotagliflozin-matching placebo tablet (identical to sotagliflozin dose 2 in appearance), once daily, before the first meal of the day
  Interventions: Drug: sotagliflozin (SAR439954); Drug: placebo
- Placebo (Placebo Comparator): Two sotagliflozin-matching placebo tablets (identical to sotagliflozin dose 2 in appearance), once daily, before the first meal of the day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Sotagliflozin dose 1; Sotagliflozin dose 2
Drug: placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo; Sotagliflozin dose 2

SUMMARY:
Primary Objective:

To demonstrate the superiority of sotagliflozin dose 1 versus placebo on hemoglobin A1c (HbA1c) reduction in Chinese patients with type 2 diabetes (T2D) who have inadequate glycemic control on diet and exercise.

Secondary Objectives:

* To compare sotagliflozin dose 1 versus placebo for change in 2-hour postprandial glucose (PPG) following a mixed meal tolerance test (MMTT), change in fasting plasma glucose (FPG), and change in body weight.
* To compare sotagliflozin dose 2 versus placebo for change in HbA1c, change in 2-hour PPG following a MMTT, change in FPG, and change in body weight.
* To compare sotagliflozin dose 2 and sotagliflozin dose 1 versus placebo for change in systolic blood pressure (SBP) for all patients, and change in SBP for patients with baseline SBP ≥130 mmHg.
* To evaluate the safety of sotagliflozin dose 2 and sotagliflozin dose 1 versus placebo.

DETAILED DESCRIPTION:
Total study duration is up to 30 weeks, including a screening period consisting of a screening phase of up to 2 weeks and a 2-week single-blind placebo run-in phase, a 24-week double-blind treatment period, and a 2-week post-treatment follow-up visit period to collect safety information.

ELIGIBILITY:
Inclusion criteria :

* Chinese patients with Type 2 Diabetes who are treated with diet and exercise only during the 12 weeks prior to screening
* Signed written informed consent.

Exclusion criteria:

* Age <18 years at the screening visit.
* Type 1 diabetes.
* Hemoglobin A1c <7% or >10% measured by the central laboratory at the screening visit.
* Fasting plasma glucose >15 mmol/L (>270 mg/dL) measured by the central laboratory at the screening visit and confirmed by a repeat test (>15 mmol/L [>270 mg/dL]) before randomization
* Body mass index (BMI) ≤20 or >45 kg/m² at the screening visit.
* Women of childbearing potential not willing to use highly effective method(s) of birth control during the study treatment period and the follow-up period, or who are unwilling or unable to be tested for pregnancy during the study.
* Previous use of any antidiabetic medication(s) for >4 months at any time or previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes).
* Previous use of any antidiabetic drug within 12 weeks prior to the screening visit.
* History of gastric surgery including history of gastric banding or inflammatory bowel disease within 3 years prior to the screening visit.
* History of diabetic ketoacidosis (DKA) or non-ketotic hyperosmolar coma within 12 weeks prior to the screening visit.
* Mean of 3 separate blood pressure measurements >180 mmHg (SBP) or >100 mmHg (diastolic blood pressure (DBP)).
* History of hypertensive emergency within 12 weeks prior to the screening visit.
* Patients with severe anemia, severe cardiovascular (CV) (including congestive heart failure New York Heart Association (NYHA) IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease or patients with short life expectancy that, according to Investigator, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of the normal (ULN) laboratory range.
* Total bilirubin >1.5 times the ULN (except in case of Gilbert's syndrome).
* Use of systemic glucocorticoids (excluding topical or ophthalmic application, nasal spray, or inhaled forms) for more than 10 consecutive days within 90 days prior to the screening visit.
* Patient who has taken other investigational drugs or prohibited therapy for this study within 12 weeks or 5 half-lives prior to the screening visit, whichever is longer.
* Pregnant (confirmed by serum pregnancy test at the screening visit) or breastfeeding women.
* Patients with severe renal disease as defined by an eGFR of <30 mL/min/1.73m² at the screening visit, based on the 4 variable Modification of Diet in Renal Disease (MDRD) equation.
* Patient unwilling or unable to perform self-monitoring of blood glucose (SMBG), complete the patient diary, or comply with study visits and other study procedures as required per protocol.
* Patients unable to consume at least 50% of the standard meal during the MMTT at baseline (Day 1, Visit 3) before randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) | Baseline to Week 24
  Absolute change from baseline to week 24 in HbA1c (for sotagliflozin dose1)

SECONDARY OUTCOMES:
Change in 2-hour postprandial glucose (PPG) following a mixed meal tolerance test (MMTT) | Baseline to Week 24
  Absolute change from baseline to week 24 in 2-hour PPG following a MMTT (for sotagliflozin dose1 and 2)
Change in fasting plasma glucose (FPG) | Baseline to Week 24
  Absolute change from baseline to week 24 in FPG (for sotagliflozin dose1 and 2)
Change in body weight | Baseline to Week 24
  Absolute change from baseline to week 24 in body weight (for sotagliflozin dose1 and 2)
Change in HbA1c | Baseline to Week 24
  Absolute change from baseline to week 24 in HbA1c (for sotagliflozin dose 2)
Change in systolic blood pressure (SBP) for all patients | Baseline to Week 12
  Absolute change from baseline to week 12 in SBP for all patients (for sotagliflozin dose1 and 2)
Change in SBP for patients with baseline SBP ≥130 mmHg | Baseline to Week 12
  Absolute change from baseline to week 12 in SBP patients with baseline SBP ≥130 mmHg (for sotagliflozin dose1 and 2)
Adverse events | Up to Week 24
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (29):
- China (29):
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560004, Beijing
  - Investigational Site Number 1560002, Beijing
  - Investigational Site Number 1560007, Changchun
  - Investigational Site Number 1560008, Changchun
  - Investigational Site Number 1560024, Chongqing
  - Investigational Site Number 1560022, Guangzhou
  - Investigational Site Number 1560033, Guangzhou
  - Investigational Site Number 1560021, Guangzhou
  - Investigational Site Number 1560029, Harbin
  - Investigational Site Number 1560009, Hohhot
  - Investigational Site Number 1560014, Huai'an
  - Investigational Site Number 1560019, Huzhou
  - Investigational Site Number 1560025, Jining
  - Investigational Site Number 1560027, Jining
  - Investigational Site Number 1560012, Luoyang
  - Investigational Site Number 1560013, Pingxiang
  - Investigational Site Number 1560034, Qingdao
  - Investigational Site Number 1560026, Qingdao
  - Investigational Site Number 1560017, Shanghai
  - Investigational Site Number 1560016, Shanghai
  - Investigational Site Number 1560006, Shijiazhuang
  - Investigational Site Number 1560005, Tianjin
  - Investigational Site Number 1560035, Wuhan
  - Investigational Site Number 1560023, Xuzhou
  - Investigational Site Number 1560028, Yinchuan
  - Investigational Site Number 1560032, Yuncheng
  - Investigational Site Number 1560015, Zhuzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org